CLINICAL TRIAL: NCT01165723
Title: A Randomised, Placebo Controlled, Double-Blind, Third Party Open, Parallel Group Study To Evaluate the Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Repeat Doses PF-04427429 Administered Intravenously To Healthy Adult Volunteers
Brief Title: A Clinical Study Evaluating The Safety And Tolerability Of PF-04427429 In Healthy Adult Volunteers. The Pharmacokinetics And Pharmacodynamics Of PF-04427429 Will Also Be Investigated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0141007
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; pharmacodynamics; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Dose 1: experimental (Experimental)
  Interventions: Biological: PF-04427429
- IV Dose 2: experimental (Experimental)
  Interventions: Biological: PF-04427429

INTERVENTIONS:
Biological: PF-04427429 — Intravenous dosing of 30mg on day 1 and one other day to be determined up to day 30
  Arms: IV Dose 1: experimental
Biological: PF-04427429 — Intravenous dosing of 30mg on day 1 and one other day to be determined up to day 30
  Arms: IV Dose 2: experimental

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-04472429 administered intravenously to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 50 years inclusive. (healthy is defined as non clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests)
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight of 50 to 100kg inclusive
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial

Exclusion Criteria:

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, genitourinary, psychiatric, neurologic or allergic disease (including drug allergies, but excluding untreated symptomatic, seasonal allergies at time of dosing)
* History of febrile illness within 5 days prior to the first dose
* A positive urine drug screen

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety (incidence/severity of adverse events and clinical laboratory abnormalities, mean change from baseline/placebo in vital signs/body temperature, mean change from baseline in 12 lead electrocardiogram parameters compared to baseline/placebo) | up to 129 days
Safety continued (categorical summary of QTcF compared to baseline between dose groups and placebo, concentration QTcF relationship, ADA responses, IV injection site reactions | up to 129 days
Pharmacokinetics (free plasma concentrations of PF-04427429 will be measured by a validated assay and non-compartmental PK parameters will be determined for each dose) | up to 129 days

SECONDARY OUTCOMES:
pharmacodynamics (free and total CGRP plasma concentration) will be measured, the PK-PD relationship between plasma PF-0447429 concentrations and free/total CGRP concentrations will be characterised | up to 129 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0141007&StudyName=A%20Clinical%20Study%20Evaluating%20The%20Safety%20And%20Tolerability%20Of%20PF-04427429%20In%20Healthy%20Adult%20Volunteers.%20The%20Pharmacokinetics%20And%20Pharmacodynamic